CLINICAL TRIAL: NCT02638753
Title: Efficacy of Education on Neurophysiology of Pain Combined to Hypnosis in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Rodrigo Rossi Nogueira Rizzo, PT, MSc Student, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNICID032016
Record Dates: First submitted 2015-12-19; First posted 2015-12-23 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Chronic Low Back Pain
Keywords: non specific chronic low back pain; education on pain neurophysiology; education on pain biology; education on pain neuroscience; hypnosis
MeSH Terms: interventions — Educational Status; Hypnosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education (Active Comparator): Patients will receive 4 sessions (1 hour each) of education on pain neurophysiology.
  Interventions: Other: education
- Education combined with hypnosis (Experimental): Patients will receive 4 sessions (1 hour each) of education on pain neurophysiology combined with hypnosis.
  Interventions: Other: education combined with hypnosis

INTERVENTIONS:
Other: education — Patients will be educated about pain neurophysiology.
  Arms: Education
Other: education combined with hypnosis — Patients will be educated about pain neurophysiology combined with hypnosis.
  Arms: Education combined with hypnosis

SUMMARY:
Although education on neurophysiology of pain improves disability, there are limited effects in pain intensity. Hypnosis is an approach that has proven useful in pain intensity and psychosocial aspects in some chronic pain conditions, but there is insufficient evidence of its contribution in patients with chronic non specific low back pain. The aim of the study is to assess the efficacy of combining education on neurophysiology of pain and hypnosis in patients with chronic non specific low back pain in pain and disability outcomes.

DETAILED DESCRIPTION:
Introduction: Education on pain neurophysiology has beneficial effects on disability and psychosocial aspects in patients with non specific chronic low back pain. However, education has limited effects in pain. Hypnosis is an approach that has proven efficient in pain intensity and psychosocial aspects in some chronic pain conditions, but there is insufficient evidence of its contribution in patients with non specific chronic low back pain.

Objectives: The aim of the study is to assess the efficacy of combining education on neurophysiology of pain and hypnosis in patients with non specific chronic low back pain in pain and disability outcomes.

Study design: randomized controlled trial with two arms and blinded evaluator. Local study: Interventions will be held at the Universidade Cidade de Sao Paulo (UNICID).

Participants: One hundred patients with chronic non specific low back pain who are on the waiting list for physical therapy care at UNICID physical therapy clinic, interested and eligible for the study will be invited to participate.

Intervention: Patients will be randomized to the education group about pain neurophysiology or to a group that combines education with hypnosis.

Measurements: Clinical outcomes will be obtained after 2 weeks and 3 months after randomization. The primary outcome will be pain intensity (measured by the numerical pain scale) and general disability (measured by the Roland-Morris questionnaire). The secondary outcome will be catastrophic thoughts (measured by PCS-Brazil), specific disability (measured by the Patient-specific function scale) and global perceived effect (measured by the Global Perceived Effect scale).

Limitations: Both the therapist and the patients will not be blinded to the intervention provided.

Hypothesis: This is the first study that will provided results achieved by education about pain neurophysiology using hypnosis in patients with chronic non specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non specific chronic low back pain, defined as pain or discomfort between the coastal margins and lower gluteal folds, with or without symptoms related to lower limbs for at least three months, of both genders, aged between 18 and 80 years and literate in Portuguese.

Exclusion Criteria:

* Patients with back pain by nerve root compromise, serious spinal pathologies (such as fracture, tumor, inflammatory and infectious diseases), cardio-respiratory and uncompensated metabolic diseases, previous back surgery , pregnancy, presence of some contraindications to exercise, and have a hearing or understanding problem that prevents the understanding of simple information.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pain Numerical Rating Scale | 2 weeks after randomization
  It is a translated and adapted scale for the Portuguese language that assesses pain intensity levels perceived by patients through a 11-point scale (ranging from 0 to 10), with 0 being classified as "no pain" and 10 "worst pain possible ". Patients will be asked to mark the level of the average pain intensity and the more intense based on the last seven days.
Roland Morris Disability Questionnaire | 2 weeks after randomization
  This questionnaire consists of 24 items describing everyday situations that patients may have difficulty in performing because of back pain. The greater the number of alternatives completed affirmatively, the greater the level of disability associated with lombar pain. Patients will be instructed to fill out the statements that actually describe their situation on the day of the interview. It's tool was already translated and adapted for the Portuguese language.

SECONDARY OUTCOMES:
The Pain Catastrophizing Scale (PCS) | 2 weeks and 3 months after randomization
  PCS is used to assess negative thoughts related to dor54. It is a self-administered questionnaire with 13 items and 3 subscales: impotence, magnification and rumination. A 5-point scale is used for each item. The score of each item is summed to define each subscale score or total score which may range from 0 to 52 points. It's tool was already translated and adapted for the Portuguese language.
The Patient-Specific Functional Scale | 2 weeks and 3 months after randomization
  We asked for the patient to identify up to 3 activities that are considered incapable of performing or presenting any difficulty. The measurement is made by Likert scale of 11 points for each activity, and the higher average score (ranging from 0 to 10 points) better is the patient's ability to make activity. It's tool was already translated and adapted for the Portuguese language.
Global Perceived Effect Scale | 2 weeks and 3 months after randomization
  It is a Likert scale of 11 points (ranging from -5 to +5) which compares the current state of the patient as the start of their symptoms. Positive scores are applied to patients who are better and negative scores apply to those who are worse off compared to the beginning of symptoms. The closer to the 5 means that the greater is the intensity perception. It's tool was already translated and adapted for the Portuguese language.
Pain Numerical Rating Scale | 3 months after randomization
  It is a translated and adapted scale for the Portuguese language that assesses pain intensity levels perceived by patients through a 11-point scale (ranging from 0 to 10), with 0 being classified as "no pain" and 10 "worst pain possible ". Patients will be asked to mark the level of the average pain intensity and the more intense based on the last seven days.
Roland Morris Disability Questionnaire | 3 months after randomization
  This questionnaire consists of 24 items describing everyday situations that patients may have difficulty in performing because of back pain. The greater the number of alternatives completed affirmatively, the greater the level of disability associated with lombar pain. Patients will be instructed to fill out the statements that actually describe their situation on the day of the interview. It's tool was already translated and adapted for the Portuguese language.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo OP Costa, PhD, Principal Investigator — Universidade Cidade de São Paulo
Locations (1):
- Universidade Cidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Airaksinen O, Brox JI, Cedraschi C, Hildebrandt J, Klaber-Moffett J, Kovacs F, Mannion AF, Reis S, Staal JB, Ursin H, Zanoli G; COST B13 Working Group on Guidelines for Chronic Low Back Pain. Chapter 4. European guidelines for the management of chronic nonspecific low back pain. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S192-300. doi: 10.1007/s00586-006-1072-1. No abstract available. PMID 16550448
- [Background] Moseley GL, Nicholas MK, Hodges PW. A randomized controlled trial of intensive neurophysiology education in chronic low back pain. Clin J Pain. 2004 Sep-Oct;20(5):324-30. doi: 10.1097/00002508-200409000-00007. PMID 15322439
- [Background] Adachi T, Fujino H, Nakae A, Mashimo T, Sasaki J. A meta-analysis of hypnosis for chronic pain problems: a comparison between hypnosis, standard care, and other psychological interventions. Int J Clin Exp Hypn. 2014;62(1):1-28. doi: 10.1080/00207144.2013.841471. PMID 24256477
- [Background] Costa LO, Maher CG, Latimer J, Ferreira PH, Ferreira ML, Pozzi GC, Freitas LM. Clinimetric testing of three self-report outcome measures for low back pain patients in Brazil: which one is the best? Spine (Phila Pa 1976). 2008 Oct 15;33(22):2459-63. doi: 10.1097/BRS.0b013e3181849dbe. PMID 18923324
- [Background] Costa LO, Maher CG, Latimer J, Ferreira PH, Pozzi GC, Ribeiro RN. Psychometric characteristics of the Brazilian-Portuguese versions of the Functional Rating Index and the Roland Morris Disability Questionnaire. Spine (Phila Pa 1976). 2007 Aug 1;32(17):1902-7. doi: 10.1097/BRS.0b013e31811eab33. PMID 17762300
- [Background] Sehn F, Chachamovich E, Vidor LP, Dall-Agnol L, de Souza IC, Torres IL, Fregni F, Caumo W. Cross-cultural adaptation and validation of the Brazilian Portuguese version of the pain catastrophizing scale. Pain Med. 2012 Nov;13(11):1425-35. doi: 10.1111/j.1526-4637.2012.01492.x. Epub 2012 Oct 4. PMID 23036076
- [Background] Chatman AB, Hyams SP, Neel JM, Binkley JM, Stratford PW, Schomberg A, Stabler M. The Patient-Specific Functional Scale: measurement properties in patients with knee dysfunction. Phys Ther. 1997 Aug;77(8):820-9. doi: 10.1093/ptj/77.8.820. PMID 9256870